CLINICAL TRIAL: NCT01204944
Title: Swiss Transplant Cohort Study
Acronym: STCS
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Bern (Other); University of Basel (Other); University of Lausanne (Other); Cantonal Hospital of St. Gallen (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Nicolas Mueller, Head, Zurich University Hospital Transplant Center, University of Zurich
Other Study IDs: 3347C0-108795/1
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2024-11

CONDITIONS: All Transplanted Individuals in Switzerland

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA Plasma PBMC
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Swiss Transplant Cohort Study is an observational prospective cohort study enrolling all patients after solid organ and stem cell transplantation since 5/2008 in Switzerland. Predefined variables are collected at defined time points. Individual samples (PBMC, plasma, DNA) will be stored for future projects. Data relevant to transplantation outcome with emphasis on immunological and infectious complications as well as psychosocial variables will be gathered.

ELIGIBILITY:
Inclusion criteria:

* All patients after organ and stem cell (planned 2009) transplantation.

Exclusion criteria:

* No informed consent given

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All transplanted indivduals in Switzerland
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2008-05; Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Outcome after transplantation | open
  Various endpoints

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Derived] Branca-Dragan S, Koller MT, Danuser B, Kunz R, Steiger J, Hug BL. Evolution of disability pension after renal transplantation: methods and results of a database linkage study of the Swiss Transplant Cohort Study and Swiss Disability Insurance. Swiss Med Wkly. 2021 Sep 23;151:w30027. doi: 10.4414/smw.2021.w30027. eCollection 2021 Sep 13. PMID 34558884
- [Derived] Krisl A, Stampf S, Hauri D, Binet I, Mueller T, Sidler D, Hadaya K, Golshayan D, Pascual M, Koller M, Dickenmann M, The Swiss Transplant Cohort Study Stcs. Immunosuppression management in renal transplant recipients with normal-immunological risk: 10-year results from the Swiss Transplant Cohort Study. Swiss Med Wkly. 2020 Dec 5;150:w20354. doi: 10.4414/smw.2020.20354. eCollection 2020 Nov 30. PMID 33277913